CLINICAL TRIAL: NCT01311219
Title: Comparison of Intramedullary Nailing, Plate Fixation, and Non-operative Treatment of Acute, Displaced, Midshaft Clavicle Fractures: a Prospective Randomized Trial
Brief Title: Study Comparing Intramedullary Nailing, Plate Fixation, and Non-operative Treatment of Clavicle Fractures
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI left institution
Sponsor: University of Missouri-Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1109438-1; NCT01307670 (obsolete NCT alias)
Record Dates: First submitted 2011-03-01; First posted 2011-03-09 (Estimated); Last update posted 2016-09-30 (Estimated); Status verified 2016-09

CONDITIONS: Clavicle Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No surgery (Active Comparator): Non-operative Treatment
  Interventions: Other: Non-operative Treatment
- Plate fixation (Active Comparator): Operative Treatment-Plate fixation
  Interventions: Procedure: Operative Treatment-Plate Fixation
- Intramedullary pinning (Active Comparator): Operative Treatment-Intramedullary Pinning
  Interventions: Procedure: Operative Treatment-Intramedullary Pinning

INTERVENTIONS:
Other: Non-operative Treatment — A figure-of-8 brace will be applied to afflicted extremity in clinic. The patient will be instructed on proper application of the brace and asked to continue wearing the brace for 2 to 6 weeks, depending on the patient's level of comfort.
  Arms: No surgery
Procedure: Operative Treatment-Plate Fixation — Plate fixation of the clavicle fracture will be performed utilizing a 3.5-mm dynamic compression plate.
  Arms: Plate fixation
Procedure: Operative Treatment-Intramedullary Pinning — Clavicle fracture will be repaired through intramedullary pinning using The Rockwood Clavicle Pin (DePuy Orthopaedics, Warsaw, IN).
  Arms: Intramedullary pinning

SUMMARY:
Patients with acute, displaced fractures of the middle third of the clavicle will be randomly assigned into either the non-operative treatment group or the operative treatment group. The operative treatment group will be randomly assigned to repair with either an intramedullary device or a plate and screws.

DETAILED DESCRIPTION:
Patients with acute, displaced fractures of the middle third of the clavicle will be randomly assigned into either the non-operative treatment group or the operative treatment group. The operative treatment group will be randomly assigned to repair with either an intramedullary device or a plate and screws. Pre-operative variables will be accounted for in detail. Operative variables including duration of surgery, length of incision, fluoroscopy times, blood loss, and quality of reduction will be recorded. Patients will be followed with regular post-operative visits in which radiographs and clinical examination will be performed. Outcome variables will include post-operative pain, time to union, union/non-union rate, return to work, return to activity, radiographic outcome, complication rates, incidence of repeat procedures, cosmesis, and functional outcome based on strength, range of motion, and scoring systems. There are five hypotheses for this study: 1) Operative treatment of acute displaced midshaft clavicle fractures will yield better patient-based functional outcomes when compared to nonoperative treatment as measured by physical assessment of strength and range of motion, standardized scoring systems and return to normal daily activities. 2) Operative treatment of acute displaced midshaft clavicle fractures will yield lower radiographically-determined nonunion rates, improved cosmesis and fewer complaints of residual pain when compared to nonoperative treatment. 3) Operative treatment of acute displaced midshaft clavicle fractures with intramedullary pinning will be more efficacious than operative treatment with plate fixation as measured by duration of surgery, length of incision, fluoroscopy time, blood loss, and quality of reduction. 4) Operative treatment of acute displaced midshaft clavicle fractures with intramedullary pinning will result in fewer complications than operative treatment with plate fixation including; nonunion rate, infection, incidence of repeat procedures, refracture rate, and hardware malfunction. 5) Operative treatment of acute displaced midshaft clavicle fractures with intramedullary pinning will yield lower radiographically-determined nonunion rates, improved cosmesis, and fewer complaints of residual pain when compared to operative treatment with plate fixation.

ELIGIBILITY:
Inclusion Criteria: All candidates with a radiographically confirmed, displaced, midshaft clavicle fracture, between the ages of 16 and 80.

-

Exclusion Criteria: Patients presenting with ipsilateral shoulder girdle injury, open fracture, pathologic fracture, or associated neurologic injury. Patients who are pregnant and therefore, unable to undergo radiologic assessment. Patients deemed incompetent to make medical decisions regarding their own health care. Patients unwilling or unable to complete postoperative evaluation at 2, 6, and 12 weeks and long term follow-up evaluation at 6 and 12 months. Prisoners who will be difficult to complete follow-up.

-

Ages: 16 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05; Primary Completion 2009-05 (Actual); Study Completion 2009-05 (Actual)

PRIMARY OUTCOMES:
Disability of the Arm, Shoulder, and Hand (DASH) | 2, 6, and 12 weeks and 6 and 12 months

SECONDARY OUTCOMES:
The Constant Pain Score | 2, 6, and 12 weeks and 6 and 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Richard A White, M.D., Principal Investigator — University of Missouri-Columbia
Locations (1):
- University of Missouri-Columbia, Columbia, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bostman O, Manninen M, Pihlajamaki H. Complications of plate fixation in fresh displaced midclavicular fractures. J Trauma. 1997 Nov;43(5):778-83. doi: 10.1097/00005373-199711000-00008. PMID 9390489
- [Background] Canadian Orthopaedic Trauma Society. Nonoperative treatment compared with plate fixation of displaced midshaft clavicular fractures. A multicenter, randomized clinical trial. J Bone Joint Surg Am. 2007 Jan;89(1):1-10. doi: 10.2106/JBJS.F.00020. PMID 17200303